CLINICAL TRIAL: NCT02284932
Title: Muscle Atrophy In Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Annie Dubé, Professionelle de recherche, Laval University
Other Study IDs: COPD-20739
Record Dates: First submitted 2014-10-08; First posted 2014-11-06 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; atrophy; muscle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — Blood sample and muscle biopsy of vastus lateralis (quadriceps)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD patients: Group : COPD patients No specific intervention for this study
  Interventions: Other: No specific intervention for this study
- Healthy controls: Group : healthy volunteers No specific intervention for this study
  Interventions: Other: No specific intervention for this study

INTERVENTIONS:
Other: No specific intervention for this study — No specific intervention for this study

SUMMARY:
Limb muscle dysfunction, characterized by atrophy and weakness, is amongst the most troublesome systemic consequences of chronic obstructive pulmonary disease (COPD) leading to poor functional status and premature mortality.

One prevailing hypothesis stipulates that the deterioration in muscle structure and function during COPD results from a spillover of inflammatory mediators from the lungs to the systemic circulation and then to the muscles.

DETAILED DESCRIPTION:
The investigators objective is to investigate the impact of COPD on key signaling pathways involved in the muscle atrophy. Moderate to severe COPD patients (FEV1 under 60% of predicted) and healthy controls will be recruited. All of the investigators patients will undergo a thorough baseline assessment in pulmonary capacity, muscle force and body composition. Blood sampling and biopsy of the quadriceps will be done. Key proteins of signaling intramuscular pathways involved in protein synthesis and degradation will be measured in the quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* male
* COPD with an FEV1 of under 60% of predicted
* non-smoker
* between 55 and 75 years old

Exclusion Criteria:

* all inflammatory disease (HIV, cancer, renal and cardiac deficiency)
* hormonal dysregulation
* inferior limb pathology
* neuromuscular pathology
* history of tobacco or alcool abuse
* oxygen dependent
* recent exacerbation (2 months) of the symptoms of COPD

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Decrease of protein degradation in muscles of wasted COPD patients | At baseline (COPD in a stable state of the disease)

SECONDARY OUTCOMES:
Increase of protein synthesis in muscles of wasted COPD patients | At baseline (COPD in a stable state of the disease)

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada